CLINICAL TRIAL: NCT00171249
Title: An Extension to a Phase II Study to Determine the Safety and Anti-Leukemic Effects of STI571 in Adult Patients With Philadelphia Chromosome Positive Leukemia Including Acute Lymphoblastic Leukemia, Acute Myeloid Leukemia, and Accelerated Phase Chronic Myeloid Leukemia
Brief Title: An Extension Study to Determine the Safety and Anti-Leukemic Effects of Imatinib Mesylate in Adult Participants With Ph+ Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571A0109E2; 2005-001381-14 (EudraCT Number)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Philadelphia Positive Chronic Myeloid Leukemia; Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia
Keywords: Chronic Myelogenous Leukemia; CML; Philadelphia Chromosome; Accelerated phase; Acute Myelogenous Leukemia; AML; Acute Lymphoblastic Leukemia; ALL; Imatinib mesylate
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Philadelphia Chromosome | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Accelerated Phase Chronic Myeloid/Myelogenous Leukemia 400 mg (Experimental): Participants with accelerated phase chronic myeloid/myelogenous leukemia received STI571 400 mg, orally, once daily, until death, the development of intolerable toxicity, or the investigator felt it was no longer in the participant's best interest to continue therapy, whichever came first.
  Interventions: Drug: STI571 400 mg
- Lymphoid Blast Crisis 400 mg (Experimental): Participants with lymphoid blast crisis received STI571 400 mg, orally, once daily, until death, the development of intolerable toxicity, or the investigator felt it was no longer in the participant's best interest to continue therapy, whichever came first.
  Interventions: Drug: STI571 400 mg
- Acute Lymphoblastic Leukemia 400 mg (Experimental): Participants with acute lymphoblastic leukemia received STI571 400 mg, orally, once daily, until death, the development of intolerable toxicity, or the investigator felt it was no longer in the participant's best interest to continue therapy, whichever came first.
  Interventions: Drug: STI571 400 mg
- Accelerated Phase Chronic Myeloid/Myelogenous Leukemia 600 mg (Experimental): Participants with accelerated phase chronic myeloid/myelogenous leukemia received STI571 600 mg, orally, once daily, until death, the development of intolerable toxicity, or the investigator felt it was no longer in the participant's best interest to continue therapy, whichever came first.
  Interventions: Drug: STI571 600 mg
- Lymphoid Blast Crisis 600 mg (Experimental): Participants with lymphoid blast crisis received STI571 600 mg, orally, once daily, until death, the development of intolerable toxicity, or the investigator felt it was no longer in the participant's best interest to continue therapy, whichever came first.
  Interventions: Drug: STI571 600 mg
- Acute Lymphoblastic Leukemia 600 mg (Experimental): Participants with acute lymphoblastic leukemia received STI571 600 mg, orally, once daily, until death, the development of intolerable toxicity, or the investigator felt it was no longer in the participant's best interest to continue therapy, whichever came first.
  Interventions: Drug: STI571 600 mg
- Acute Myeloid/Myelogenous Leukemia 600 mg (Experimental): Participants with acute myeloid/myelogenous leukemia received STI571 600 mg, orally, once daily, until death, the development of intolerable toxicity, or the investigator felt it was no longer in the participant's best interest to continue therapy, whichever came first.
  Interventions: Drug: STI571 600 mg

INTERVENTIONS:
Drug: STI571 400 mg — STI571 capsules and tablets
  Other Names: Imatinib mesylate; Glivec®; GleevecTM
  Arms: Accelerated Phase Chronic Myeloid/Myelogenous Leukemia 400 mg; Acute Lymphoblastic Leukemia 400 mg; Lymphoid Blast Crisis 400 mg
Drug: STI571 600 mg — STI571 capsules and tablets
  Other Names: Imatinib mesylate; Glivec®; GleevecTM
  Arms: Accelerated Phase Chronic Myeloid/Myelogenous Leukemia 600 mg; Acute Lymphoblastic Leukemia 600 mg; Acute Myeloid/Myelogenous Leukemia 600 mg; Lymphoid Blast Crisis 600 mg

SUMMARY:
The objectives of Part 1 of the study were:

* To determine the rate of hematologic response (HR) lasting ≥4 weeks in participants with Philadelphia chromosome-positive (Ph+) chronic myeloid leukemia (CML) in the accelerated phase (AP).
* To evaluate duration of HR, overall survival, cytogenetic response (CyR), time to blast crisis in CML participants in the AP, improvement of symptomatic parameters, tolerability and safety of STI571 treatment.

The objective of the extension (Part 2) was:

-To enable participants to have access to study drug and continue study treatment and to decrease data collection to include only overall survival and serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants, aged ≥18 years, with a histologically confirmed diagnosis of Ph+ leukemia of one of the following types:

  * Accelerated phase chronic myeloid/myelogenous leukemia (CML).
  * Acute lymphoid/lymphoblastic leukemia (ALL) or acute myeloid/myelogenous leukemia (AML) in first or subsequent relapse after either standard chemotherapy, autologous or allogeneic bone marrow transplantation, or high-dose treatment with peripheral blood stem cell support, or
  * ALL or AML refractory to standard chemotherapy (no complete remission achieved after two courses of conventional induction chemotherapy).
  * Lymphoid blastic phase of CML in first or subsequent relapse or refractory to standard chemotherapy.
* With serum serum glutamate oxaloacetate transaminase (aspartate aminotransferase) and serum glutamate pyruvate transaminase (alanine aminotransferase) not more than 3 x upper limit of normal (ULN) (or not more than 5xULN if clinically suspected leukemic involvement of the liver), serum creatinine concentration not more than 2xULN, and total serum bilirubin level not more than 3xULN (bilirubin limit was 1.5xULN before protocol amendment 1)

Exclusion Criteria:

* Participants who had an Eastern Cooperative Oncology Group (ECOG) performance status score ≥3.
* Participants with known leukemic involvement of the central nervous system (CNS).
* Participants who had received treatment with any of the following agents: interferon-alpha within 48 hours, hydroxyurea within 24 hours, homoharringtonine within 14 days, low-dose, moderate dose or high dose cytosine arabinoside within 7, 14 or 28 days respectively, 6-mercaptopurine, vinca alkaloids or steroids within 7 days, anthracyclines, mitoxantrone, etoposide, methotrexate, cyclophosphamide within 21 days, or busulfan within 6 weeks.
* Participants who had undergone hematopoietic stem cell transplantation within six weeks of Day 1, or who had not achieved full hematopoietic recovery following the transplant.
* Participants with grade 3/4 cardiac disease or any serious, concomitant, medical condition.
* Participants with a history of non-compliance to medical regimens or who were considered potentially unreliable.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 293 (Actual)
Dates: Start 1999-08-09 (Actual); Primary Completion 2013-09-23 (Actual); Study Completion 2013-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- United States (4):
  - Dana Faber Cancer Institute, Boston, Massachusetts
  - New York Presbyterian Hospital, New York, New York
  - Oregon Health & Sciences University, Portland, Oregon
  - MD Anderson Cancer Center, University of Texas, Houston, Texas
- France (2):
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Poitiers
- Germany (4):
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Mannheim
- Novartis Investigative Site, Monza, Italy
- Novartis Investigative Site, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in this study at 14 investigative sites in France, Germany, Italy, United Kingdom, Switzerland and United States from August 9, 1999 to September 23, 2013.
Pre-assignment Details: On July 31, 2002, the core study was completed and 76 participants on study medication were enrolled to the extension protocol #1 (E1), and as of July 31, 2004, 42 participants were still on treatment and were enrolled in a further extension protocol #2 (E2).
Period: Overall Study
Arm/Group | Accelerated Phase Chronic Myeloid/Myelogenous Leukemia 400 mg | Lymphoid Blast Crisis 400 mg | Acute Lymphoblastic Leukemia 400 mg | Accelerated Phase Chronic Myeloid/Myelogenous Leukemia 600 mg | Lymphoid Blast Crisis 600 mg | Acute Lymphoblastic Leukemia 600 mg | Acute Myeloid/Myelogenous Leukemia 600 mg
Started | 77 | 5 | 5 | 158 | 3 | 43 | 2
Completed Part 1 | 50 | 0 | 1 | 125 | 2 | 6 | 0
Completed | 1 | 0 | 0 | 6 | 0 | 0 | 0
Not Completed | 76 | 5 | 5 | 152 | 3 | 43 | 2
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 6 | 0 | 0 | 0
Not completed — Unsatisfactory Therapeutic Effect | 44 | 3 | 5 | 70 | 3 | 31 | 1
Not completed — Death | 7 | 1 | 0 | 4 | 0 | 3 | 1
Not completed — Other | 10 | 0 | 0 | 43 | 0 | 2 | 0
Not completed — No Longer Requires Study Drug | 4 | 0 | 0 | 3 | 0 | 5 | 0
Not completed — Administrative Problems | 1 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 1 | 0 | 15 | 0 | 2 | 0
Not completed — Lost to Follow-up | 5 | 0 | 0 | 9 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) population consisted of all enrolled participants. Baseline characteristics were collected and reported together for each disease and dose groups (Accelerated Phase Chronic Myeloid/Myelogenous Leukemia 400 mg or 600 mg, Lymphoid Blast Crisis 400 mg or 600 mg, Acute Lymphoblastic Leukemia 400 mg or 600 mg, and Acute Myeloid/Myelogenous Leukemia 600 mg) of participants, as pre-specified in the protocol.
Groups:
- STI571: Participants received STI571 400/600 mg, orally, once daily, until death, the development of intolerable toxicity, or the investigator felt it was no longer in the participant's best interest to continue therapy, whichever came first.
  Note- Data is reported with data that is available. No additional data tables were found that could provide results 'per arm' , therefore a summary arm has been reported.
Arm/Group | STI571
Number analyzed (Participants) | 293
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (12.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146
  Male | 147

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Hematologic Response in Accelerated Phase Chronic Myeloid/Myelogenous Leukemia
Description: Hematologic response was evaluated from hematology measurements in the peripheral blood (PB) and bone marrow (BM) and assessments of extramedullary leukemic involvement (EMD) at physical examination. Response was defined as complete hematologic remission (CHR), no evidence of leukemia (NEL), or return to chronic phase (RTC).
Time Frame: Up to 3 years after start of treatment
Population: ITT population consisted of all enrolled participants. The data for this outcome measure was collected and analyzed in participants who belonged to the disease group of Accelerated Phase Chronic Myeloid/Myelogenous Leukemia 400 mg or 600 mg only, as pre-specified in the protocol. The other three acute leukemia disease groups were exploratory only.
  Data is reported with data that is available. No additional data tables were found that could provide results with arms broken down any further.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Accelerated Phase Chronic Myeloid/Myelogenous Leukemia 400 mg | Accelerated Phase Chronic Myeloid/Myelogenous Leukemia 600 mg
Number analyzed (Participants) | 77 | 158
percentage of participants | 64.9 [53.2 to 75.5] | 74.7 [67.2 to 81.3]

2. Secondary Outcome: Percentage of Participants With Cytogenetic Response in Accelerated Phase Chronic Myeloid/Myelogenous Leukemia
Description: Bone marrow (BM) cytogenetic analysis was required at baseline, after 12 weeks (visit 22) and after 24 weeks (visit 28) to evaluate Ph chromosome positivity. In several participants, this was also done after 4 and 8 weeks. Based on the percentage of Philadelphia chromosome positive (Ph+) cells = (positive cells/examined cells)x100, at each BM assessment the cytogenetic response was classified as: Complete, 0% Ph+ cells; Partial, >0 - 35% Ph+ cells; Minor, >35 - 65% Ph+ cells; Minimal, >65 - 95% Ph+ cells; None, >95% Ph+ cells; Not done: <20 metaphases were examined and/or response could not be assigned. Cytogenetic response was defined as confirmed complete or partial response. A BM sample was considered as assessable for cytogenetic response only if it contained ≥20 metaphases. However, an assessment of partial response was retained in a sample with <20 metaphases when it was immediately preceded or followed by a complete or partial response in another sample with ≥20 metaphases.
Time Frame: Up to 3 years after start of treatment
Population: ITT population consists of all enrolled participants. The data for this outcome measure was collected and analyzed in participants who belonged to the disease group of Accelerated Phase Chronic Myeloid/Myelogenous Leukemia 400 mg or 600 mg only, as pre-specified in the protocol. The other three acute leukemia disease groups were exploratory only.
  Data is reported with data that is available. No additional data tables were found that could provide results with arms broken down any further.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Accelerated Phase Chronic Myeloid/Myelogenous Leukemia 400 mg | Accelerated Phase Chronic Myeloid/Myelogenous Leukemia 600 mg
Number analyzed (Participants) | 77 | 158
percentage of participants | 14.3 [7.4 to 24.1] | 24.7 [18.2 to 32.2]

3. Secondary Outcome: Time to Response in Participants With Accelerated Phase Chronic Myeloid/Myelogenous Leukemia
Description: Time to response was defined for all participants as the time until first documented response (which was confirmed ≥4 weeks later).
Time Frame: Up to 3 years after start of treatment
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Accelerated Phase Chronic Myeloid/Myelogenous Leukemia 400 mg | Accelerated Phase Chronic Myeloid/Myelogenous Leukemia 600 mg
Number analyzed (Participants) | 77 | 158
months
  Hematologic response: number analyzed (Participants) | 50 | 118
  Hematologic response | 0.95 [0.95 to 1.1] | 0.99 [0.99 to 1]
  Cytogenetic response: number analyzed (Participants) | 15 | 49
  Cytogenetic response | 2.83 [1.9 to 5.6] | 2.96 [2.8 to 5.5]

4. Secondary Outcome: Duration of Response in Participants With Accelerated Phase Chronic Myeloid/Myelogenous Leukemia
Description: Duration of response was defined as the time between first documented response (which was confirmed ≥4 weeks later) and the earliest date of the following: loss of response (when any of the criteria for response were no longer fulfilled); progression to blast crisis (≥30% blasts in peripheral blood or bone marrow, extramedullary involvement other than liver/spleen enlargement); discontinuation due to adverse event, laboratory abnormality, unsatisfactory therapeutic effect or death.
Time Frame: Up to 3 years after start of treatment
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Accelerated Phase Chronic Myeloid/Myelogenous Leukemia 400 mg | Accelerated Phase Chronic Myeloid/Myelogenous Leukemia 600 mg
Number analyzed (Participants) | 77 | 158
months
  Hematologic response: number analyzed (Participants) | 50 | 118
  Hematologic response | 16.46 [10.4 to 27.4] | 28.81 [25.7 to NA] — Upper limit of 95% CI was not estimable due to censored data
  Cytogenetic response: number analyzed (Participants) | 15 | 49
  Cytogenetic response | 26.28 [6.6 to NA] — Upper limit of 95% CI was not estimable due to censored data | 27.63 [15.9 to NA] — Upper limit of 95% CI was not estimable due to censored data

5. Secondary Outcome: Time to Progression to Blast Crisis in Participants With Accelerated Phase Chronic Myeloid/Myelogenous Leukemia
Description: Progression to blast crisis was defined as ≥30% blasts in peripheral blood or bone marrow or as extramedullary involvement other than liver or spleen enlargement.
Time Frame: Up to 3 years after start of treatment
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Accelerated Phase Chronic Myeloid/Myelogenous Leukemia 400 mg | Accelerated Phase Chronic Myeloid/Myelogenous Leukemia 600 mg
Number analyzed (Participants) | 77 | 158
months | 9.95 [6.6 to 14.4] | 25.13 [18.1 to 29.8]

6. Secondary Outcome: Overall Survival by Disease
Description: To evaluate overall survival, all participants were followed after the last dose of study drug every month for the first three months and thereafter every three months until death. Overall survival was calculated for all participants as the time between start of treatment and death due to any reason. The time was censored at the date of last contact for participants who discontinued treatment and were in survival follow-up. For participants without survival follow-up information, the time was censored at last available visit/treatment date.
Time Frame: 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, and 156 months after start of treatment
Population: ITT population consisted of all enrolled participants. The data for this outcome measure was collected and analyzed in participants by disease groups.
  Data is reported with data that is available. No additional data tables were found that could provide results with arms broken down any further.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Accelerated Phase Chronic Myeloid/Myelogenous Leukemia: Participants with accelerated phase chronic myeloid/myelogenous leukemia received STI571 400/600 mg, orally, once daily, until death, the development of intolerable toxicity, or the investigator felt it was no longer in the participant's best interest to continue therapy, whichever came first.
- Lymphoid Blast Crisis: Participants with lymphoid blast crisis received STI571 400/600 mg, orally, once daily, until death, the development of intolerable toxicity, or the investigator felt it was no longer in the participant's best interest to continue therapy, whichever came first.
- Acute Lymphoid Leukemia: Participants with acute lymphoid leukemia received STI571 400/600 mg, orally, once daily, until death, the development of intolerable toxicity, or the investigator felt it was no longer in the participant's best interest to continue therapy, whichever came first.
- Acute Myeloid/Myelogenous Leukemia: Participants with acute myeloid/myelogenous leukemia received STI571 600 mg, orally, once daily, until death, the development of intolerable toxicity, or the investigator felt it was no longer in the participant's best interest to continue therapy, whichever came first.
Arm/Group | Accelerated Phase Chronic Myeloid/Myelogenous Leukemia | Lymphoid Blast Crisis | Acute Lymphoid Leukemia | Acute Myeloid/Myelogenous Leukemia
Number analyzed (Participants) | 235 | 8 | 48 | 2
percentage of participants
  12 months | 74.4 [68.3 to 79.5] | 12.5 [0.7 to 42.3] | 10.4 [3.8 to 20.9] | 0 [0 to 0]
  24 months | 58.8 [52.2 to 64.8] | 0 [0 to 0] | 8.3 [2.7 to 18.2] | 0 [0 to 0]
  36 months | 48 [41.4 to 54.2] | 0 [0 to 0] | 8.3 [2.7 to 18.2] | 0 [0 to 0]
  48 months | 39.9 [33.5 to 46.2] | 0 [0 to 0] | 8.3 [2.7 to 18.2] | 0 [0 to 0]
  60 months | 32.2 [26.1 to 38.4] | 0 [0 to 0] | 8.3 [2.7 to 18.2] | 0 [0 to 0]
  72 months | 26.3 [20.6 to 32.3] | 0 [0 to 0] | 8.3 [2.7 to 18.2] | 0 [0 to 0]
  84 months | 24.1 [18.6 to 30.1] | 0 [0 to 0] | 8.3 [2.7 to 18.2] | 0 [0 to 0]
  96 months | 21.9 [16.5 to 27.8] | 0 [0 to 0] | 5.6 [1.2 to 15.2] | 0 [0 to 0]
  108 months | 20.6 [15.3 to 26.4] | 0 [0 to 0] | 5.6 [1.2 to 15.2] | 0 [0 to 0]
  120 months | 20.6 [15.3 to 26.4] | 0 [0 to 0] | 5.6 [1.2 to 15.2] | 0 [0 to 0]
  132 months | 18.9 [13.6 to 24.8] | 0 [0 to 0] | 5.6 [1.2 to 15.2] | 0 [0 to 0]
  144 months | 18.9 [13.6 to 24.8] | 0 [0 to 0] | 5.6 [1.2 to 15.2] | 0 [0 to 0]
  156 months | 18.9 [13.6 to 24.8] | 0 [0 to 0] | 5.6 [1.2 to 15.2] | 0 [0 to 0]

7. Secondary Outcome: Overall Survival by Dose in Participants With Accelerated Phase Chronic Myeloid/Myelogenous Leukemia
Description: as for outcome 6
Time Frame: 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, and 132 months after start of treatment
Population: ITT population consisted of all enrolled participants. The overall survival was calculated as per initial dose (400 mg or 600 mg) only for participants with Accelerated Phase Chronic Myeloid/Myelogenous Leukemia, as pre-specified in the protocol.
  Data is reported with data that is available. No additional data tables were found that could provide results with arms broken down any further.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Accelerated Phase Chronic Myeloid/Myelogenous Leukemia 400 mg | Accelerated Phase Chronic Myeloid/Myelogenous Leukemia 600 mg
Number analyzed (Participants) | 77 | 158
percentage of participants
  12 months | 64.5 [52.6 to 74.1] | 79.1 [71.9 to 84.7]
  24 months | 44.3 [32.9 to 55.1] | 65.7 [57.7 to 72.6]
  36 months | 34.9 [24.4 to 45.7] | 54.2 [46.0 to 61.6]
  48 months | 28.0 [18.4 to 38.5] | 45.6 [37.6 to 53.2]
  60 months | 23.7 [14.7 to 33.9] | 36.2 [28.6 to 43.9]
  72 months | 18.6 [10.5 to 28.5] | 29.9 [22.6 to 37.5]
  84 months | 15.2 [7.8 to 24.8] | 28.3 [21.2 to 35.9]
  96 months | 11.8 [5.4 to 21.0] | 26.6 [19.6 to 34.2]
  108 months | 11.8 [5.4 to 21.0] | 24.8 [17.9 to 32.3]
  120 months | 11.8 [5.4 to 21.0] | 24.8 [17.9 to 32.3]
  132 months | 11.8 [5.4 to 21.0] | 22.3 [15.4 to 29.9]

ADVERSE EVENTS:
Time Frame: Up to approximately 14 years
Description: AEs were not collected separately for each disease and dose groups of participants. The data has been reported as originally produced by the team at the time of reporting. We have exhausted all efforts to locate additional data; therefore, no additional data is available to report or modify what has previously been reported. No other non-serious AEs were collected during extension phase within clinical database.
Arm/Group | STI571
Serious Adverse Events (participants affected / at risk) | 20/293
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | STI571 (N=293)
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Dementia Alzheimer's type (Nervous system disorders) | 1
Death (General disorders) | 2 — Sudden death
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Atypical mycobacterial infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.